CLINICAL TRIAL: NCT07228338
Title: Muscarinic Agonist Modulation of Memory Processing Oscillatory Activity
Brief Title: Cholinergic Enhancement of Theta
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Bradley Lega, Professor - Neurological Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU20250602
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Epilepsy; Seizures; Cognitive Impairment, Mild; Memory Disorder; Memory Loss
Keywords: oscillatory changest; cholinergic agonist; muscarinic agonist
MeSH Terms: conditions — Epilepsy; Seizures; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Patients are randomized to COBENFY or placebo by the pharmacy. Both researchers and patients are blinded to which session receives pharmaceutical versus placebo administration. Each of the patients receive COBENFY or placebo on Day 1 and Day 2 before completing tasks at to evaluate effects on episodic memory processes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- COBENFY KarXT (50/20 mg) (Experimental): Subjects will receive a dose of COBENFY KarXT (50/20 mg). Approximately 2 hours minutes after administration, the participant will then complete an episodic memory task session. If the patient completed the sham session already, this session will take place minimum of 24 hours following the initial session, or at least four half-lives after the first session.
  Interventions: Drug: COBENFY KarXT (50/20 mg)
- Placebo (Placebo Comparator): Subjects will receive a placebo. Approximately 2 hours minutes after administration, the participant will then complete an episodic memory task session. If the patient completed the COBENFY KarXT session already, this session will take place minimum of 24 hours following the initial session, or at least four half-lives after the first session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COBENFY KarXT (50/20 mg) — Patient receives a dose of COBENFY KarXT (50/20 mg) 2 hours prior to episodic memory task.
  Arms: COBENFY KarXT (50/20 mg)
Drug: Placebo — Patient receives a dose of placebo 2 hours prior to episodic memory task.
  Arms: Placebo

SUMMARY:
The goal of this study is to learn about the effects of Cobenfy KarXT (xanomeline and trospium chloride) on episodic memory processing, including specific effects on areas of the brain involved in memory and changes it may have on brain activity. The investigators will do this by testing epileptic patients who are already undergoing intracranial surgery for seizure monitoring, and measuring the activity from the brain areas being assessed.

The main questions it aims to answer are 1) whether Cobenfy KarXT changes memory activity based on its agonist effect on muscarinic receptors and acetylcholine, and 2) what the nature of these brain activity changes are. This work builds on previous experiments evaluating cholinergic antagonists.

Participants will complete two treatment arms. One of these will be with the drug, and the other will be with a placebo pill, so that the participants are unaware which session the actual drug has been received. Patients will complete a verbal serial recall and/or associative recognition task each of the two days. An anesthesiologist or patient nurse will administer either the drug or the placebo at a critical point which addresses both of the research questions.

Researchers will compare the brain activity between the two treatment arms to determine what brain activity changes, and whether there is an additional behavioral effect on memory.

DETAILED DESCRIPTION:
Patient Identification: The study team plans to recruit adult patients who are undergoing invasive electroencephalographic (EEG) monitoring as part of standard clinical procedure for the treatment of pharmacologically resistant epilepsy at UT Southwestern. Patients are identified from the pool of patients presented at the epilepsy management conference and approached when they present to the clinic for evaluation for seizure surgery. Patients are screened by a coordinator as well as anesthesiologist on the study team for contraindications which make them ineligible for receiving the drug.

Study procedures: Participation takes place only during the time that the electrodes are surgically in place. Active participation will end when the electrodes are removed. Tasks described below will be administered by key personnel on the study. The data will be de-identified and converted to signal data for processing and analysis. Study personnel, excluding the PI (aka 'experimenters') will perform analysis.

Once patients are in the epilepsy monitoring unit (EMU), subjects will be randomized to receive either a dose of 50 mg/20 mg orally BID of xanomeline and trospium chloride (COBENFY) or placebo pill. Approximately 2 hours after administration, the participant will complete an episodic memory task session. At least 24 hours following the first session (at least four half-lives after the first session), the participant will receive the alternative agent not given the first day. For example, if the patient received COBENFY the first day, they would receive the placebo the second day, and vice versa. They will then complete an additional episodic memory task session 2 hours after administration.

Day 1: Randomized to receive either COBENFY or placebo (sham); Complete episodic memory task session Day 2: Receives alternate agent from day 1; Completes episodic memory task session

Participant will not know whether Cobenfy KarXT is being administered, or if he/she receives the placebo. Researchers will be blind to this until after patient has completed both sessions. The randomization will be generated by the pharmacy using a psuedorandomizer.

The participant's attending nurse will administer Cobenfy KarXT and/or placebo 2 hours prior to the test.

Physiologic Monitoring: Patients in the epilepsy monitoring undergo EKG and pulse oxygen monitoring in addition to seizure monitoring electrodes at all times as part of routine care and this will not be interrupted during the study period. There is a certified epilepsy monitoring team available should the cholinergic effects enhance seizures. A board-certified anesthesiologist with specialist practice in neuroanesthesia will be immediately available within the hospital to respond with any other concerns. In our previous experiments using cholinergic modulation (antagonism), there have not been any adverse events. Specifically, there has not been an impact on seizure activity. While we do not anticipate an effect of Cobenfy KarXT on seizure activity, we note that all patients are located in the EMU environment with 2:1 nursing ratios and immediately available protocols for interventions if seizures occur.

Overview of Memory Testing: Episodic memory tasks in our lab typically last 30-75 minutes provided patient does not request a break during the task. There is no physical risk to participants from cognitive tasks. Participants may stop and resume each task whenever they need a break. Participants for this protocol would need to wait at least 24 hours/six half-lives following completion of one of the testing sessions prior to completing the second, regardless of whether administration of either placebo or Cobenfy KarXT occurred. The cognitive tasks will cause patients to incur no additional medical or surgical risk; rather patients often report the game-like testing protocols provide relief from the boredom of awaiting seizures. Within each session, patients may request breaks to avoid fatigue. Testing may also be paused or interrupted for any health-care-related needs. The research team will attend to the comfort of all participants, who may discontinue the testing at any time, without repercussions.

Episodic Memory Tasks: Patients will participate in verbal memory tasks, such as lists of specific words to be recalled freely or in a serial order. such lists are comprised of words or nameable pictures. A computer controls stimulus presentation and records participants' response of words or word order. Each list is followed by a brief distractor task consisting of a simple addition or subtraction problem prior to recall. This end-of-list distracter task serves to reduce the large advantage accorded to end-of-list items during recall, or recency effect. There are approximately 10-12 words or items in one list. Participants are then given the opportunity to place these words in the order they recall them. Their responses are digitally recorded by the computer and anonymously stored for later analysis. This paradigm cannot specifically address questions regarding differences on encoding versus retrieval, so patients may be also be given other types of verbal memory tasks, such as recognition paradigms of associative recognition, or other verbal tasks that will be able to parse out such aspects of episodic memory.

Collection of iEEG data: Patients included in the study undergo the acquisition of EEG data for clinical purposes by clinicians, using a computerized EEG collection system. In this study, we will copy these data, strip them of any confidential information, and analyze the raw traces of EEG. Synchronization of the experimental computer with the iEEG signals is accomplished by sending an optically isolated pulse to an input on the EEG recording system. This train of pulses enables the iEEG record to synchronize itself with the testing computer, in standard fashion for this work.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years, all races/ethnicities, and both genders are eligible.
2. Candidates for pre-operative evaluation using stereo intracranial electrodes and admission to the Epilepsy Monitoring Unit (EMU) as determined independently by the patient's treating physician as part of the patient's routine medical care.
3. Able to read, understand, and provide written, dated informed consent prior to screening.
4. In good general health, aside from a history of epilepsy, as ascertained by medical history, physical examination (PE), clinical laboratory evaluations, and ECG.

Exclusion Criteria:

1. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results according to the study physician.
2. Female that is pregnant, breastfeeding, or has a positive pregnancy test at screening or baseline. We note that pregnant patients are excluded from undergoing iEEG.
3. Hepatic impairment (moderate or severe).
4. Renal impairment (moderate or severe).
5. Clinically significant bladder outlet obstruction or incomplete bladder emptying, such as patients with prostatic hyperplasia (BPH), diabetic cystopathy, pre-existing urinary retention.
6. History of hypersensitivity to COBENFY or trospium chloride (angioedema risks).
7. Untreated narrow-angle glaucoma.
8. Biliary Disease (symptomatic gallstones, gallbladder disorders, pancreatitis).
9. Strong Inhibitors of CYP2D6 such as fluoxetine, paroxetine, bupropion, terbinafine.
10. Sensitive Substrates of CYP3A4 such as buspirone, eletriptan.
11. Narrow Therapeutic Index Substrates of P-glycoprotein such as digoxin, colchicine, apixaban.
12. Drugs Eliminated by Active Tubular Secretion.
13. Antimuscarinic Drugs such as diphenhydramine, benztropine, oxybutynin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the Free recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta power and oscillatory changes. Other changes, such as phase amplitude coupling, may also be considered.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the Free recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta power and oscillatory changes. Other changes, such as phase amplitude coupling, may also be considered.
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the serial recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily thetapower and oscillatory changes. Other changes, such as phase amplitude coupling, may also be considered.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the serial recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta power and oscillatory changes. Other changes, such as phase amplitude coupling, may also be considered.
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the associative recognition memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta power and oscillatory changes. Other changes, such as phase amplitude coupling, may also be considered.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the associative recognition memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta power and oscillatory changes. Other changes, such as phase amplitude coupling, may also be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C Lega, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No